CLINICAL TRIAL: NCT00965835
Title: Amyloid Plaque and Tangle Imaging in Alzheimer's Disease and Down Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Linda Nelson, Ph.D., Emerita, Professor of Psychiatry and Biobehavioral Sciences, Semel Institute
Other Study IDs: IA0166; 1R21AG030681-01A2 (NIH)
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Down Syndrome; Alzheimer's Disease
Keywords: PET Scan
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DS: Those with Down syndrome
- Non-DS: Healthy controls

SUMMARY:
The purpose of this study is to develop small molecule radio-labeled probes of beta-amyloid, to be used with positron emission tomography (PET) for early detection and treatment monitoring of Alzheimer disease (AD). The study hypothesis is that PET imaging of small molecule probes, in the form of novel fluorescent dyes with radioactive labels, will demonstrate cerebral patterns in patients with AD that are distinct from those of age-matched persons who are cognitively intact.

DETAILED DESCRIPTION:
This is a naturalistic study in which clinical evaluations and brain scans will be performed on 20 people with Down syndrome (DS) as well as 20 healthy controls across a range of ages. Participants will receive comprehensive clinical and neuropsychological assessments. PET and MRI scans will be performed at baseline and after two years of follow up. All participants will have blood drawn for APOE genotyping during their baseline evaluations. The intellectual range of participants with DS will be restricted to IQ scores of 45 to 60 (moderate range) to reduce variability, particularly due to extreme low levels of intellectual ability.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* No significant cerebrovascular disease - modified Ischemic Score of < 4
* Adequate visual and auditory acuity to allow neuropsychological testing
* Screening laboratory tests and ECG without significant abnormalities that might interfere with the study

Additional Inclusion Criteria for Controls

* MMSE score between 24 and 30 (unless < 8 years of educational achievement)
* The following medications are allowed if stable for > 1 month: antidepressants (without anticholinergic effects) if not currently depressed and no history of major depression for 2 years; estrogen replacement therapy; thyroid replacement therapy as long as individual is euthyroid; antihypertensives that do not influence cognitive function

Additional Inclusion Criteria for Individuals with Down syndrome

* Family member or caregiver available; caregiver relationship 2 years or longer
* Karyotype DX of trisomy or translocation DS Mosaic form of Down syndrome
* English-speaking

Exclusion Criteria:

* Evidence of neurological or other physical illness that could produce cognitive deterioration; volunteers with a history of TIAs, carotid bruits, or lacunes on MRI scan will be excluded
* Parkinson's Disease
* History of myocardial infarction within the previous year or unstable cardiac disease
* Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100), history of significant liver disease, clinically significant pulmonary disease, diabetes, or cancer
* Major psychiatric disorders, such as bipolar disorder or schizophrenia
* Medicines that could influence psychometric test results
* Use of any of the following drugs: centrally active beta-blockers, narcotics, clonidine, anti-Parkinsonian medications, benzodiazepines, systemic corticosteroids, medications with significant cholinergic or anticholinergic effects, anti-convulsants, or warfarin
* Current diagnosis or history of alcoholism or drug dependence
* Evidence of untreated depression or untreated anxiety
* Use of any investigational drugs within the previous month or longer, depending on drug half-life
* Contraindication for MRI scan (e.g., metal in body, claustrophobia)
* Diagnosis of possible or probable AD or any other dementia (e.g., vascular, Lewy body, frontotemporal) or MCI

Additional Exclusion Criteria for Individuals with Down syndrome

* Mosaic form of Down syndrome
* History of clinically significant neurological disorder or disease and Psychiatric diagnosis or treatment within 3 months prior to screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals will be identified and recruited using IRB approved flyers distributed to treating clinicians, caregivers from Board and Care homes, sheltered workshop administrators (where potential participants are employed), and representatives of County Regional Centers (primary evaluation and treatment centers for developmentally delayed individuals).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Nelson, PhD, Principal Investigator — Semel Institute, UCLA
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] Nelson LD, Scheibel KE, Ringman JM, Sayre JW. An experimental approach to detecting dementia in Down syndrome: a paradigm for Alzheimer's disease. Brain Cogn. 2007 Jun;64(1):92-103. doi: 10.1016/j.bandc.2007.01.003. Epub 2007 Mar 26. PMID 17383786
- [Background] Nelson LD, Orme D, Osann K, Lott IT. Neurological changes and emotional functioning in adults with Down Syndrome. J Intellect Disabil Res. 2001 Oct;45(Pt 5):450-6. doi: 10.1046/j.1365-2788.2001.00379.x. PMID 11679050
- [Background] Small GW, Kepe V, Ercoli LM, Siddarth P, Bookheimer SY, Miller KJ, Lavretsky H, Burggren AC, Cole GM, Vinters HV, Thompson PM, Huang SC, Satyamurthy N, Phelps ME, Barrio JR. PET of brain amyloid and tau in mild cognitive impairment. N Engl J Med. 2006 Dec 21;355(25):2652-63. doi: 10.1056/NEJMoa054625. PMID 17182990
- [Background] Small GW, Siddarth P, Burggren AC, Kepe V, Ercoli LM, Miller KJ, Lavretsky H, Thompson PM, Cole GM, Huang SC, Phelps ME, Bookheimer SY, Barrio JR. Influence of cognitive status, age, and APOE-4 genetic risk on brain FDDNP positron-emission tomography imaging in persons without dementia. Arch Gen Psychiatry. 2009 Jan;66(1):81-7. doi: 10.1001/archgenpsychiatry.2008.516. PMID 19124691